CLINICAL TRIAL: NCT00404521
Title: A Phase I Single-institution, Open-label, Dose-escalating, Clinical and Pharmacokinetic Study of PM02734 Administered Every 3 Weeks, Intravenously, Over 30 Minutes, to Subjects With Advanced Malignant Solid Tumors.
Brief Title: A Phase I Study of PM02734 in Subjects With Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low rate recruitment
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM2734-A-001-05
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Solid Tumors
Keywords: Tumor; PM02734; PharmaMar
MeSH Terms: conditions — Neoplasms | interventions — elisidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: PM02734

INTERVENTIONS:
Drug: PM02734 — Administered every 3 weeks, intravenously, over 30 minutes

SUMMARY:
Phase I single-institution, open-label, dose-escalating, clinical and pharmacokinetic study. The purpose is to determine the safety, tolerability and to identify the dose limiting toxicities(DLT) and recommended dose (RD) of PM02734 administered every 3 weeks, intravenously, over 30 minutes to subjects with advanced malignant solid tumors.

DETAILED DESCRIPTION:
Phase I single-institution, open-label, dose-escalating, clinical and pharmacokinetic study. The purpose is to determine the safety, tolerability and to identify the dose limiting toxicities(DLT) and recommended dose (RD) of PM02734 administered every 3 weeks, intravenously, over 30 minutes to subjects with advanced malignant solid tumors. Secondary objectives are to determine preliminary Pharmacokinetics of PM02734, to explore the relationships between pharmacokinetics and pharmacodynamics. To evaluate the preliminary pharmacokinetics/pharmacodynamics correlation and to evaluate the preliminary antitumor activity of PM02734. The trial will be conducted in compliance with the protocol, GCP and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the subject obtained before any study-specific procedure.
2. Histologically or cytologically confirmed malignant solid tumor.
3. Subjects with malignancies for which no standard therapy would reasonably be expected to result in cure or palliation.
4. Age ≥ 18 years.
5. Subject with measurable or non-measurable disease using the RECIST criteria (only subjects with measurable disease are allowed to enter the expanded cohort).
6. Recovery from any drug-related adverse event derived from previous treatment, excluding alopecia and NCI-CTCAE grade 1 symptomatic peripheral neuropathy.
7. Laboratory values within 7 days prior to first infusion:

   * Platelet count ≥ 100 x109/L , hemoglobin > 9 g/dL and absolute neutrophil count (ANC) ≥ 1.5 x109/L.
   * Alkaline phosphatase ≤ 2.5 x the upper limit of normality (ULN) (< 5 x ULN in case of extensive bone metastases).
   * Aspartate aminotransferase (AST): ≤ 2.5 x ULN (<5 x ULN in case of extensive liver metastases).
   * Alanine aminotransferase (ALT): ≤ 2.5 x ULN (<5 x ULN in case of extensive liver metastases).
   * Total bilirubin:1.5 ≤ ULN, unless due to Gilbert's syndrome.
   * Creatinine: ≤ ULN, or measured creatinine clearance: ≥ 60 mL/min without significant proteinuria (>250 mg/m2 /day)
   * Albumin ≥ 2.5 g/dL.
   * Partial thromboplastin time ≤ 1.1 x ULN
   * INR ≤ 1.1
8. Performance status (ECOG) ≤ 2 .
9. Life expectancy ≥ 3 months.
10. Left ventricular ejection fraction (LVEF) within normal limits.
11. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both men and women must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment. Acceptable methods of contraception include complete abstinence, IUD, oral contraceptive, subdermal implant and double barrier (condom with a contraceptive sponge or contraceptive suppository).

Exclusion Criteria:

1. Prior therapy with PM02734.
2. Pregnant or lactating women.
3. Less than 4 weeks from radiation therapy (8 weeks in case of extensive prior radiotherapy) or last dose of hormonal therapy, biological therapy or chemotherapy (6 weeks in case of nitrosourea, mitomycin C, or high-dose chemotherapy).
4. Evidence of progressive CNS metastases or any symptomatic brain or leptomeningeal metastases.
5. Evidence of extensive liver metastases ( more than 5 hepatic nodules and some of them greater than 5 cm in diameter)
6. Other relevant diseases or adverse clinical conditions:

   * Increased cardiac risk: congestive heart failure or unstable angor pectoris or arrhythmia requiring treatment or uncontrolled arterial hypertension or myocardial infarction within 12 months before inclusion in the study.
   * History of significant neurological or psychiatric disorders.
   * Active infection.
   * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
   * Significant non-neoplastic renal disease.
   * Immunocompromised subjects, including subjects known to be infected by human immunodeficiency virus (HIV).
   * Uncontrolled endocrine diseases (e.g. diabetes mellitus, hypothyroidism or hyperthyroidism, adrenal disorder) (i.e. requiring relevant changes in medication within the last month or hospital admission within the last 3 months).
   * Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study.
7. Limitation of the subject's ability to comply with the treatment or to follow-up at a participating protocol. Subjects registered on this trial must be treated and followed at a participating center.
8. Treatment with ongoing anti-coagulation.
9. Treatment with any investigational product in the 30 days period prior to the first infusion.
10. Known hypersensitivity to any of the components of the drug product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, dose limiting toxicities (DLT) and recommended dose (RD) of PM02734 | Along the study

SECONDARY OUTCOMES:
To determine preliminary pharmacokinetics, to explore relationships between pharmacokinetics/pharmacodynamics correlation and to evaluate preliminary antitumor activity of PM02734 | Along the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ratain, MD, Principal Investigator — Cancer Research Centerr, University of Chicago Hospital
Locations (1):
- Cancer Research Center. University of Chicago Hospitals, Chicago, Illinois, United States